CLINICAL TRIAL: NCT02445105
Title: Mobilizing Community Systems to Engage Families in Early Autism Spectrum Disorder (ASD) Detection & Services
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Florida State University (Other)
Collaborators: Emory University (Other); Weill Medical College of Cornell University (Other); Drexel University (Other); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Amy M. Wetherby, Distinguished Research Professor, Florida State University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: MH104423; 1R01MH104423-01 (NIH)
Record Dates: First submitted 2015-04-01; First posted 2015-05-15 (Estimated); Last update posted 2022-07-13 (Actual); Status verified 2022-07

CONDITIONS: Autism Spectrum Disorder
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Autism Navigator Enhanced Practice (Active Comparator): A 6-hour training will be provided to community service providers with the Autism Navigator for Primary Care professional development course and use of a web-based platform that includes an automated communication and autism screening and monthly electronic monitoring.
  Interventions: Behavioral: Autism Navigator Enhanced Practice
- Family Engagement plus Autism Navigator (Experimental): A 6-hour training will be provided to community service providers on the use of Motivational Interviewing, an evidence-based counseling method to improve engagement of families who are ambivalent about screening or intervention for their toddler, in addition to Autism Navigator Enhanced Practice.
  Interventions: Behavioral: Family Engagement plus Autism Navigator

INTERVENTIONS:
Behavioral: Autism Navigator Enhanced Practice — Community service providers will receive training in Autism Navigator for Primary Care, a 6-hour online professional development course with extensive video illustration of the early signs of autism in toddlers, collaborating with families, developmental milestones, screening and referral practices, and early intervention basics. This web-based platform includes an automated screening for communication delay and autism, an automated monthly electronic monitoring, and digital tools for families to address practical obstacles to screening toddlers 9-18 months of age and referral to early intervention.
  Arms: Autism Navigator Enhanced Practice
Behavioral: Family Engagement plus Autism Navigator — Community service providers will receive a 6-hour training on the use of Motivational Interviewing, an evidence-based counseling method to improve engagement of families who are ambivalent about screening or intervention for their toddler. Community service providers will also receive a 6-hour training with the Autism Navigator for Primary Care professional development course and use of the web-based platform that includes an automated communication and autism screening and monthly electronic monitoring to address practical obstacles to screening toddlers 9-18 months of age and referral to early intervention.
  Arms: Family Engagement plus Autism Navigator

SUMMARY:
This multisite study will compare the effectiveness of universal screening by 3 community service systems using Autism Navigator, a highly interactive web platform that includes an automated screening tool, information about autism for families, and a professional development course on the early signs of autism and effective evidence-based practice with extensive video footage to rapidly build the capacity for early detection. The investigators will also conduct a multisite pragmatic randomized clinical trial to test the effectiveness of an evidence-based Family Engagement Intervention compared to Autism Navigator Enhanced Practice implemented by the 3 community service systems with children who have a positive autism screen to increase the number of children who are screened, referred for evaluation, receive a diagnosis, and receive community-based EI between 18-27 months of age. This study will impact family engagement in community screening and diagnosis by demonstrating the effectiveness of brief manualized engagement interventions. Findings will advance science by providing researchers with a method for recruiting a community sample, allowing for research at younger ages, which could accelerate science.

DETAILED DESCRIPTION:
The American Academy of Pediatrics recommends screening all children for autism spectrum disorder (ASD) at 18 and 24 months because research indicates that earlier intervention maximizes children's outcomes. The earliest signs of ASD are delays in social communication milestones that appear in the first 2 years and yet most children are not diagnosed until 4-5 years of age. Underserved families are identified even later and significantly underrepresented in intervention research. It is vitally important to mobilize community service systems to impact family engagement throughout the process of screening, evaluation, and early intervention (EI) and to support linkages to public community-based EI in order to address health disparities. This collaborative investigation of 4 universities aims to document the effectiveness of an online automated universal screen for communication delay and autism initially at 18 months of age and decision rule for referral to an ASD evaluation, and to study an evidence-based intervention to increase family engagement and expedite receipt of screening, diagnosis, eligibility for EI, and EI services. The study will focus on the youngest age when ASD can be detected reliably, which is 18 months, and compare the effectiveness of screening and referral by 3 different community service systems: 1) primary care including private and public health care agencies and federally qualified health centers; 2) federal programs such as Women, Infants, and Children (WIC) Food and Nutrition Service and Early Head Start; and 3) the National Black Church Initiative (NBCI). Using the Autism Navigator web-based platform the investigators will expand their capacity for universal ASD screening and referral for diagnosis and determining eligibility by EI providers through the public Individuals with Disabilities Education Act (IDEA) Part C system for children birth to 3 years of age. Innovative web-based technology will be integrated at multiple levels- as the basis for an interactive professional development course to enable these community service systems to efficiently learn about autism and implement a universal broadband and autism-specific screening with seamless automation that links to electronic health records and provides families with web-based tools about autism. This multidisciplinary research team will conduct a multisite pragmatic randomized clinical trial to test the effectiveness of an evidence-based Family Engagement Intervention plus Autism Navigator compared to Autism Navigator Enhanced Practice alone. The investigators will also conduct an exploratory study to test strategies to improve uptake of evidence-based intervention by community-based EI providers through the Part C system. This protocol has the potential to lower the age of screening for ASD to 18 months, which will have important implications for earlier access to intervention and improving ASD service systems and be ready for immediate and rapid implementation in community settings across the US. Findings will advance science by providing researchers with a method for recruiting a population-based sample, allowing for research at younger ages, which could accelerate genetic, neuroscience, and intervention research, and lead to transformative changes to community healthcare delivery.

ELIGIBILITY:
Inclusion Criteria:

1. Community service providers will be recruited from the specific catchment areas of the 4 sites in Florida, Georgia, New York, and Pennsylvania from 3 different community service systems:

   1. primary care including private, public, and military health care agencies and federally qualified health centers;
   2. federal programs including Women, Infants, and Children (WIC) Food and Nutrition Service, Early Head Start, and other social programs supporting low-income families; and
   3. the National Black Church Initiative (NBCI) and other religious networks serving minorities.
2. Children are screened between 9 and 18 months of age by these community service providers who have agreed to be in this study and their families.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10857 (Actual)
Dates: Start 2015-12; Primary Completion 2021-06 (Actual); Study Completion 2021-06 (Actual)

PRIMARY OUTCOMES:
Number of children screened by community service provider | 9 to 36 months of age
  This is a tally of the number of children screened by each provider and then summed.
Child age at screening by community service provider | 9 to 36 months of age
  This is the age of the child at the time of screening in months.
Child age at referral for evaluation by community service provider | 9 to 36 months of age
  This is the age that the child is referred by the provider for an evaluation in months.
Child age at entry into intervention | 9 to 36 months of age
  This is the age that the child enters and begins early intervention in months.

SECONDARY OUTCOMES:
Child autism symptoms measured with the Autism Diagnostic Observation Schedule | when child is 27 and 36 months of age
  Autism symptoms measured with the Autism Diagnostic Observation Schedule
Child developmental level measured with the Mullen Scales of Early Learning | when child is 27 and 36 months of age
  Developmental level measured with the Mullen Scales of Early Learning
Child adaptive behavior measured with the Vineland Adaptive Behavior Scales | when child is 27 and 36 months of age
  Adaptive behavior measured with the Vineland Adaptive Behavior Scales
Family measure of resources measured with Family Resource Scale completed by parent | when child is 27 and 36 months of age
  Family Resource Scale completed by parent
Family measure of stress measured with Parenting Stress Index completed by parent | when child is 27 and 36 months of age
  Parenting Stress Index completed by parent
Family measure of access to community activities measured with Home and Community Activities Survey completed by parent | when child is 27 and 36 months of age
  Home and Community Activities Survey completed by parent to rate how often the parent and child participate in 30 different activities and how important each activity is.

CONTACTS AND LOCATIONS:
Overall Officials: Amy M Wetherby, PhD, Principal Investigator — Florida State University
Locations (4):
- United States (4):
  - Florida State University, Tallahassee, Florida
  - Emory University, Atlanta, Georgia
  - Weill Cornell Medical College, White Plains, New York
  - Drexel University, Philadelphia, Pennsylvania